CLINICAL TRIAL: NCT01240044
Title: Study of Respiratory Therapy and Newborn Pain That Made a Comparison Between Physiotherapeutical Techniques
Brief Title: Respiratory Therapy and Newborn Pain: Comparison Between Techniques
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of the State of Santa Catarina (Other)
Responsible Party: Principal Investigator, Camila Isabel Santos Schivinski, Dr., University of the State of Santa Catarina
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PTNB 2010
Record Dates: First submitted 2010-11-12; First posted 2010-11-15 (Estimated); Last update posted 2013-06-19 (Estimated); Status verified 2010-10

CONDITIONS: Newborn Pain; Respiratory Therapy Techniques
Keywords: Newborn Pain; Respiratory Physiotherapy; Neonatal intensive care unit
MeSH Terms: interventions — Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Control Group (No Intervention): In this group the newborns remained at rest 20 minutes and receive no intervention of respiratory therapy.
- Physical Therapy (Experimental): In this group the newborns are submitted to the mechanical vibrator.
  Interventions: Procedure: Physical Therapy
- Thoracoabdominal rebalancing (Experimental): In this group the newborns receive the thoracoabdominal rebalancing.
  Interventions: Procedure: Thoracoabdominal rebalancing

INTERVENTIONS:
Procedure: Thoracoabdominal rebalancing — In this group the infants received four handlings thoracoabdominal rebalancing, in order: 1) 5min support thoracoabdominal, in which the therapist leaned one hand on the lower chest and upper abdomen of the newborn, with some of its fingers on the ribs, pulling them gently down and keeping them in that position during inspiration, 2) more than 5 minutes of abdominal support, carried by hand in the lower abdomen of the newborn, applying light pressure during inspiration enough to be beaten by the diaphragm of the newborn and not to increase the use of accessory muscles of inspiration, 3) 5min support ileo-costal, by a slight manual pressure of the physiotherapist on the lateral chest and abdomen of the newborn, maintained throughout inspiration and 4) finally ran up 5min ginga thoracic maneuver slight manual pressure on the lower chest of newborns, directing the costal movement during expiration, now an then the other hemithorax.
  Arms: Thoracoabdominal rebalancing
Procedure: Physical Therapy — In this group the newborns were first submitted to the mechanical vibrator applied over a diaper, on the chest of newborns for 5 min, as follows: 1min 1min right hemithorax and the left hemithorax, both previously, followed 30 seconds in the lateral aspect of each hemithorax; more than 1min in each hemithorax in the posterior region. The mechanical vibrator was performed subsequent to manual chest compression, using light hand pressure on the chest of newborns, respecting the compliance of the chest. The chest compression was applied for 2min 2min in the right hemithorax and left-sided chest, above, and 1 minute on each side, another 2 minutes on the back of each hemithorax, totaling 10 minutes of compression. Next to chest compression, mechanical vibration was applied for 5 min in the same topographical sequence described.
  Arms: Physical Therapy

SUMMARY:
This study intend to assess the pain intensity of newborns in neonatal intensive care unit (NICU) undergoing different techniques of respiratory therapy and compare these procedures. A randomized controlled clinical trial and blind trial with newborns admitted to NICU. The babies were categorized according to gestational age , age, weight, diagnosis, support and signs of respiratory distress. Then, they were allocated by lot to come from one of 3 groups: G1 - control, G2 - undergoing physical therapy; G3 - received the thoracoabdominal rebalancing. Each newborn received just one physical therapy session in that they were assessed before one of the three procedures (T1), immediately after (T2) and after 15 minutes (T3). This evaluation found cardiorespiratory parameters (oxygen saturation, heart and respiratory rate) and three specific scales for pain assessment (NIPS, NFCS and PIPP). The hypothesis is that newborns hospitalized in intensive care unit did not show pain when undergoing respiratory therapy.

ELIGIBILITY:
Inclusion Criteria:

* Newborns up to 28 days with any weight and gestational age in ventilatory support or oxygen therapy and clinical indication for Physical Therapy.

Exclusion Criteria:

* Newborns with contraindication of respiratory therapy, those that had problems during any of the study procedures and changes in those suffering from respiratory support or oxygen therapy during data collection.
* If there was failure to collect any of the parameters for evaluating the newborn also was no longer part of the sample.

Ages: 1 Day to 28 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2010-07; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Changes in cardiorespiratory parameters | Immediately after intervention and 15 minutes after the end of the intervention
Pain Scales (NIPS, PIPP, NFCS) | Immediately after intervention and 15 minutes after the end of the intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Maternidade Carmela Dutra Hospital, Florianópolis, Santa Catarina, Brazil